CLINICAL TRIAL: NCT02507141
Title: Reflectance Confocal Microscopy of Oral Cancers in Vivo: a Preliminary Trial Comparing Intra-oral Imaging With Pathology
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-128
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma (SCC) of the Oral Cavity
Keywords: Reflectance Confocal Microscopy; 15-128
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples of tissue from tumor and margin

GROUPS / COHORTS (1):
- SCC of the oral cavity scheduled for surgery: The patients will be imaged for testing the feasibility of intra-oral imaging. Images will be compared to and evaluated against the corresponding pathology that is routinely prepared during surgery.
  Interventions: Device: Reflectance Confocal Microscopy

INTERVENTIONS:
Device: Reflectance Confocal Microscopy — Reflectance Confocal Microscopy imaging will be performed during surgery. The imaging procedure is expected to last no more than 15-20 minutes. The approach will be essentially similar to the imaging of skin cancer on patients, which is routinely performed in our Dermatology Service.

SUMMARY:
The purpose of this study is to get images (pictures) of oral lesions, which occur inside the mouth, before the patient's surgery using a special camera. These pictures will be used in our research to evaluate a new technology that uses a laser and takes pictures of the microscopic structure of tissue. The technology is called "reflectance confocal microscopy." We would like to compare what the camera sees to biopsies (pathology) of the same area. We will evaluate the pictures obtained from the patient to determine whether this technology may be useful in the future. We hope this technology can be used as a tool for early diagnosis of oral cancers and for guiding surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven oral SCC who are scheduled to undergo surgery in the MSK Head and Neck Service.
* Ability to sign informed consent.
* Age ≥ 18 years.

Exclusion Criteria:

* Cancer located on a site that may not be convenient or accessible for imaging with the current version of the RCM device (gingivobuccal region, back of the oral cavity, back of the tongue, floor of the mouth, deep under the tongue, etc.).
* Inability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects in the Head and Neck Service will be identified by a member of the patient's treatment team, the protocol investigator, or a member of the research team at Memorial Sloan Kettering Cancer Center (MSK).
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2015-07-21 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Reflectance Confocal Microscopy (RCM) images | 1 year
  Each set of images and the corresponding pathology will be evaluated by the study pathologist for the presence or absence of oral SCC. All images will be evaluated as a group. First, the pathologist will review the RCM images for each imaging site and will determine the presence/absence of tumor. Next, the pathologist will review the corresponding histopathologic material for the presence/absence of tumor. If there is discordance in the evaluations, the pathologist will re-evaluate the RCM images with the corresponding pathology, in a side-by-side manner, to highlight any features that may assist in the RCM evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Snehal Patel, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Basking Ridge (consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (consent only), Middletown, New Jersey
  - Memorial Sloan Kettering West Harrison (consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (consent only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/